CLINICAL TRIAL: NCT03326687
Title: Pairing Word Retrieval and Physical Endurance Tasks to Treat Anomia
Brief Title: Pairing Word Retrieval and Physical Endurance Tasks to Treat Anomia in People With Aphasia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient personnel
Sponsor: University of Nebraska Lincoln (Other)
Collaborators: Quality Living, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17337
Record Dates: First submitted 2017-10-20; First posted 2017-10-31 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Aphasia
Keywords: Language; Anomia; Therapy
MeSH Terms: conditions — Aphasia; Language; Anomia

STUDY DESIGN:
Intervention Model Description: All participants will receive both the isolated and combined treatments in an ABAB or BABA order of phases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment ABAB (Experimental): Participants will receive anomia treatment in isolation and will perform a physical endurance task in isolation during A phases. They will receive anomia treatment in combination with performing a physical endurance task during B phases.
  Interventions: Behavioral: Treatment ABAB
- Treatment BABA (Experimental): Participants will receive anomia treatment in isolation and will perform a physical endurance task in isolation during A phases. They will receive anomia treatment in combination with performing a physical endurance task during B phases.
  Interventions: Behavioral: Treatment BABA

INTERVENTIONS:
Behavioral: Treatment ABAB — Participants will perform the phases in the ABAB order.
  Arms: Treatment ABAB
Behavioral: Treatment BABA — Participants will perform the phases in the BABA order.
  Arms: Treatment BABA

SUMMARY:
Many individuals have difficulty with word retrieval, also called anomia, following cerebrovascular accident (CVA). These difficulties impede effective communication in everyday conversations and can negatively impact the resumption of pre-injury activities. Even after rehabilitation specifically targeting these areas, many individuals report persistent difficulties with anomia. Additionally, most individuals report that these difficulties worsen when distracted, fatigued, or when attempting to divide attention between tasks. Given that everyday activities frequently require efficient communication when attention is divided (e.g., walking and talking), it is important to investigate viable interventions to improve these skills.

Recovery from CVA and resumption of pre-injury activities is best supported by rehabilitation interventions that are functional and directly related to the tasks individuals aim to resume. For example, a therapy task requiring an individual to generate a grocery list and then go to a grocery store to acquire the items on the list has a greater impact on recovery for the underlying language and cognitive skills than a series of generic language and cognition tasks completed in a therapy room. In addition to this, interventions that incorporate dual-task practices tend to have better outcomes than more traditional single-task practices.

The aim of this study is to compare the effectiveness of pairing word retrieval tasks with physical endurance tasks versus presenting them in isolation. Additionally, this study will investigate whether improvements in word retrieval and physical endurance generalize to the functional, everyday task of holding a conversation while walking. The researchers hypothesize that participants will perform better on word retrieval tasks after participating in dual language and physical tasks than after participating in language tasks presented in isolation.

DETAILED DESCRIPTION:
All data collection will occur at Quality Living (QLI).

The researchers will administer a set of standardized assessments prior to initiating the intervention program to determine eligibility for study participation as well as to gather descriptive information about the language abilities of participants. Assessments will include the Western Aphasia Battery - Revised and the Boston Naming Test. In addition to performing language assessments, participants will respond to demographic and injury-related questions and will identify preferred topics of conversation. The researchers will obtain information about each participant's physical status by referring to the physical therapy assessments and associated documentation completed by a QLI physical therapist shortly after the individual's arrival at QLI.

Intervention will occur five days per week and will take place during participants' regularly scheduled speech therapy sessions. Two intervention sessions will occur daily, one held in the morning and the second held in the afternoon. Depending on the activities performed on a given day, the total time devoted to intervention sessions will be 10 to 30 minutes (i.e., 5 to 15 minutes per session).

During each intervention session, the researchers will measure performance on one or more of the following tasks: (a) five trials of generative naming given a unique category and one-minute response period per trial, (b) distance traveled using an exercise machine for five minutes, (c) generative naming given unique categories and one-minute response periods and distance traveled using an exercise machine when performing both tasks simultaneously for five minutes, (d) number of words generated in five minutes in response to conversational topic prompts, (e) distance traveled when walking for five minutes, and (f) number of words generated in response to conversational topic prompts and distance traveled when walking when performing both tasks simultaneously for five minutes. The first three measures comprise intervention tasks, and the remaining three are generalization measures.

Intervention and generalization sessions will follow an overlapping ABAB or BABA format, with the first day of each phase being an overlap day. Participants will be randomly assigned to begin the intervention either with an A or B phase. On overlap days, the researchers will collect measures on all six intervention and generalization activities, with three being performed during a fifteen-minute morning session and three being performed during a fifteen-minute afternoon session. For participants in the A phase, the researchers will collect measures two times daily for each of the subsequent four days on the generative naming and exercise machine activities performed as independent tasks; for participants in the B phase, the researchers will collect measures two times daily for each of the subsequent four days on the generative naming and exercise machine activities performed as simultaneous tasks. A phase sessions will last ten minutes each, and B phase sessions will last five minutes each. The cycle of A and B phases will repeat throughout a participants inpatient stay at QLI. A QLI physical therapist will be present to monitor safety during performance of physical activities. The researchers will audio record all generative naming and conversational discourse activities for later analysis.

Participants will only perform naming, discourse, and physical endurance tasks that are included as part of their routine speech-language therapy and physical therapy sessions. However, completion of the physical endurance tasks will not occur during the participants' physical therapy sessions; instead, they will occur during speech-language therapy sessions. The naming and discourse tasks will also occur during the participants' speech-language therapy sessions.

ELIGIBILITY:
Inclusion Criteria:

* Have acquired brain injury due to left cerebrovascular accident (CVA)
* Be older than 19 years of age
* Speak English as a native language
* Be less than 3 months post-left CVA at the time of participation initiation
* Use natural speech as a primary means of communicating
* Have hearing adequate for conversational speech
* Have mild to moderate deficits in word retrieval and physical endurance as a result of left CVA
* Be currently receiving treatment services at Quality Living for CVA-related deficits

Exclusion Criteria:

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
Number of words named in a category | One or two times daily until discharge from the facility (up to 24 weeks).
  The researcher will provide a participant with a category label. The participants will name as many words as he/she can in that category within a one-minute time period. The researcher will tally the total number of unique and category-appropriate words named.

SECONDARY OUTCOMES:
Distance traveled (in feet) while using an exercise machine | One or two times daily until discharge from the facility (up to 24 weeks).
  The participant will walk on an exercise machine. The distance (measured in feet) will be measured during a five-minute time period.
Number of words generated during discourse | Two times per week until discharge from the facility (up to 24 weeks).
  The researcher will give each participant a verbal prompt to initiate and sustain a five-minute discourse about one of the topics he/she selected prior to beginning the intervention. The conversational interaction will be audio recorded for later analysis and tallying of the number of words generated by the participant.
Distance traveled (in feet) while walking | Two times per week until discharge from the facility (up to 24 weeks).
  The participant will walk a specified route inside the Quality Living facility. The distance (measured in feet) will be measured during a five-minute time period.

CONTACTS AND LOCATIONS:
Overall Officials: Karen A Hux, PhD, Principal Investigator — University of Nebraska Lincoln; Carly R Dinnes, MA, Principal Investigator — University of Nebraska Lincoln
Locations (1):
- Quality Living, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
The researchers do not plan to share IPD because of the potential for violation of participants' privacy and confidentiality is too great given the participant pool.